CLINICAL TRIAL: NCT02538744
Title: Complementary Combination Therapy for Cocaine Dependence
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Christopher Verrico, Associate Professor, Psychiatry Research, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H36362
Record Dates: First submitted 2015-08-25; First posted 2015-09-02 (Estimated); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Cocaine Dependence
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Doxazosin; Modafinil; Cocaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo (Placebo Comparator): placebo po 1x/day from day -12 through 4
  Interventions: Drug: Doxazosin; Drug: Modafinil; Drug: cocaine; Drug: Placebo
- doxazosin 8 mg (Active Comparator): day -12 through -9: Doxazosin 1 mg po 1x/day day -8 through -5: Doxazosin 2 mg po 1x/day day -4 through -1: Doxazosin 4 mg po 1x/day day 1 through 4: Doxazosin 8 mg po 1x/day
  Interventions: Drug: Doxazosin; Drug: Modafinil; Drug: cocaine; Drug: Placebo

INTERVENTIONS:
Drug: Doxazosin — Participants will be randomized into two groups: placebo and doxazosin 8 mg/d. The doxazosin dose will be increased every 4 days over 11 days, starting with 1mg on the first study day and and ending with 8mg 11 days later. Participants will receive one capsule daily that will contain either placebo or doxazosin.
Drug: Modafinil — After titrating doxazosin to the target dose, study procedures will be completed three times, once during treatment with each dose of modafinil (0 [placebo], 200, and 300 mg/d), in pseudo-random order such that 200 mg precedes 300 mg).
Drug: cocaine — On the 5th day of study medication treatment participants will receive non-contingent doses of cocaine (placebo, 20, 40 mg, IV) and participate in cocaine self-administration sessions.
Drug: Placebo

SUMMARY:
The investigators will assess the impact of treatment with doxazosin and modafinil, alone and in combination, on the subjective and reinforcing effects of cocaine in non-treatment-seeking, cocaine-dependent volunteers. The investigators will use a hybrid design in which participants will be randomized into two groups: placebo and doxazosin 8 mg/d. They will remain in their assigned group for the duration of the study. After titrating doxazosin to the target dose, study procedures will be completed three times, once during treatment with each dose of modafinil (0, 200, and 300 mg/d), in pseudo-random order such that 200 mg precedes 300 mg).

DETAILED DESCRIPTION:
During a screening session participants will provide buccal swab for genetics testing, as preliminary data shows that effects of cocaine and of doxazosin are impacted significantly by the genotype at ADRA1A, in that those with the CC genotype respond robustly to both cocaine and doxazosin whereas those with the CT genotype do not. Participants will be enrolled regardless of genotype, though the investigators plan to retrospectively exclude those with the rare TT genotype.

During screening, the investigators will collect participants' demographic and medical histories, conduct a physical exam, and record an ECG. A trained assistant will administer the MINI to collect diagnostic data. The investigators will draw blood and for CBC and a comprehensive metabolic panel including electrolytes, liver function tests (total bilirubin, ALT, AST, and alkaline phosphatase) and renal function tests (creatinine and BUN).

All applicants for study participation will receive counseling as part of their participation, and will be advised that treatment for drug abuse is indicated and available. Applicants not participating in the study will receive treatment referral information as appropriate. At completion of their participation, study subjects will again be advised that treatment is indicated and available, and will be given treatment referral information and assistance.

General Procedures Participants will report to the research commons three-times-weekly during the 11 day doxazosin titration period. They will be allowed to miss up to 3 visits but will be discontinued if they miss more that 3 visits. At the initial screening visit, restrictions on use of alcohol, drugs of abuse, and medications will be reviewed. All subjects will be required to sign a written statement that they will abstain from all psychostimulants throughout the duration of their participation in the trial.

After determining that volunteers meet inclusion and exclusion criteria, participants will receive screening doses of cocaine (0, 20, 40 mg, IV, constrained such that 20 mg precedes 40 mg). To be retained in the study participants must report a change in ratings of "high" of at least 20 points from before to following the 40 mg dose.

Remaining participants will be randomized into the two treatment groups (placebo and doxazosin 8 mg/d). Doxazosin will be titrated to the target dose over 11 days to minimize side-effects. Participants will complete the doxazosin titration phase of the study as outpatients because doxazosin alone is known to be safe when combined with cocaine. Participants will report to research commons every 4 days. The titration schedule is attached in Table 2.

The investigators will use standard riboflavin labeling to monitor treatment adherence throughout the study. Riboflavin (25mg) will be encapsulated with the study medication and adherence will be monitored by measuring riboflavin in urine using quantitative fluorescence 39,40. Because riboflavin is contained in many vitamin preparations, positive riboflavin tests may not truly reflect adherence to study medication treatment. To confirm adherence, the investigators will add 15 mg acetazolamide (ACZ) to the doxazosin capsules. ACZ will be included in doxazosin study medication from the beginning of the study until day 6 when capsules not containing ACZ will be substituted. The team will continue monitoring urine for several days after day 6 to characterize how long it takes for ACZ to become undetectable.

Participants must test cocaine negative on day 1 or they will be discontinued from the study, though they may reenter later if the investigators agree. After dose titration investigators will initiate treatment with the target doses of study medications. As shown below in Table 3 (attached), participants remain in their original doxazosin treatment group for the duration of the study (the two groups are listed to emphasize this point). Participants will complete non-contingent cocaine dosing and cocaine self-administration procedures three times, once during treatment with each dose of modafinil. Non-contingent dosing and self-administration will be done on the same day, with non-contingent dosing occuring in the am and self-administration in the pm. One treatment order is illustrated (0, 200, 300 mg/d), but in practice the order in which participants receive the three modafinil doses (placebo, 200 mg/d, and 300 mg/d) will be randomized.

Participants will be followed as outpatients for most of the study. They report to the clinic about every 4 days as shown in Table 3 for observed dosing and urine testing for adherence monitoring. Participants must test cocaine-negative on days 1, 4, 9, and 14 to remain in the study. This is so that participants are not enrolled in the study or admitted to research commons with unknown amounts of cocaine in their bodies.

Participants will take three capsules daily at 7:00 am. The capsules will contain placebo, doxazosin 8 mg, or modafinil 200 or 300 mg, depending on their randomization group and modafinil dose. On the 4th day of study medication treatment they will be admitted to research commons to ensure that procedures the following day occur under fairly standard conditions. On the 5th day of study medication treatment they will receive non-contingent doses of cocaine and participate in cocaine self-administration sessions. After completing these study activities, modafinil will be discontinued and there will be a modafinil wash-out period of 4 days during which time they will continue to take their assigned dose of doxazosin. They will then complete the study procedures during treatment with their next assigned modafinil dose. This will be repeated until participants have completed the study three times, once at each modafinil dose. As noted above, participants remain in their original doxazosin treatment group and participants continue to receive their assigned doxazosin dose throughout the study.

Daily activities for the non-contingent cocaine dosing days are shown in Table 4 and daily activities for the cocaine self-administration days are shown in Table 5 (see section S for all tables). Non-contingent doses of cocaine (placebo, 20, 40 mg, IV) will be administered at hourly intervals in random order. The following day there will be two self-administration sessions. In one session doses placebo saline will be available and in another session doses of 20 mg cocaine will be available with the order counterbalanced across participants. At the beginning of each session participants will receive a sample of the drug available in that session, saline or cocaine. The will then make a series of 10 choices between receiving the drug available in that session and monetary alternatives of increasing value. The value of the money choices will increase over the 10 choices: $.05, $.05, $.05, $.05, $1, $4, $7, $10, $13, $16. Choices will occur at 15 min intervals. The investigators have previously found that this arrangement produces choice behavior that reflects the magnitude of reinforcing effects and that is sensitive to pharmacologic manipulation.

Criteria for Withholding Cocaine Cocaine will not be administered if there are behavioral manifestations of cocaine toxicity (agitation, psychosis, inability to cooperate with study procedures), though this has not been observed with the small doses of cocaine administered in human laboratory studies. To ensure that subjects will not be at risk from cocaine, the resting pulse must be less than 90 bpm and the blood pressure must be less than 150 mmHg systolic and less than 90 mmHg diastolic.

Criteria for Participant Discontinuation:

1. Positive urine drug screen or breath test indicating illicit use of abused drugs not delivered as part of this protocol
2. Inability to comply with study procedures
3. Have exaggerated response to cocaine (5 min or more of systolic BP greater than 180 mmHg, diastolic BP greater than 120 mmHg, or heart rate greater than [(220 - age) × 0.85] bpm).

Cocaine Administration and Medical Monitoring Participants will remain seated during experimental sessions except for brief visits to the lavatory. An IV will be placed for cocaine dosing. On days involving non-contingent cocaine dosing, after first confirming that vital signs are within allowed limits, the physician will administer solution by slow IV push. An ACLS-certified physician will be present from 15 min before drug administration until at least 1 hour after drug administration. The physician will be available in house and on pager for at least 4 hours after drug administration. Heart rate will be measured using continuous ECG from 15 min prior to cocaine or placebo dosing until 1 hour after dosing. Blood pressure will be assessed at frequent intervals from 15 min prior to cocaine or placebo dosing assessment for 1 hour after dosing or until baseline levels reached.

On days involving choice sessions, an IV will be placed and patient-controlled analgesia (PCA) pump will be loaded with saline or 20mg cocaine doses depending on the session. Participants will receive one non-contingent sample dose of the drug available that session. Participants will then have 10 opportunities to choose between receiving repeated doses of the drug available that session (which will be the same as the sample dose) or receiving monetary alternatives of increasing value ($.05, $.05, $.05, $.05, $1, $4, $7, $10, $13, $16). Choices will begin 15 min after the sample dose and subsequent choices will be available at 15 min intervals.

Cocaine dosing will be delayed if necessary due to elevated cardiovascular indices based on the stopping criteria above. Investigators selected the 15 min inter-dose interval for use in the self-administration sessions based on published data showing that this arrangement is safe and yields interpretable data 44. Heart rate will be monitored continuously and blood pressure will be measured prior to dosing at 15 min intervals until 45 min after the final cocaine dose. The physician will halt cocaine administration if stopping criteria are met.

Assessments Substance Use Inventory (SUI). This instrument collects data on the type, frequency, and amounts of drugs used, as well as routes of administration. Participants will complete this measure during screening before each of the inpatient episodes. DSM-IV Diagnosis. The MINI will be administered during the initial screening and serves to determine whether the participant meets the DSM-IV criteria for drug dependence and to rule out any major psychiatric disorders (e.g., affective disorders, schizophrenia). Data from the SUI can be used to augment the ability of the MINI to determine if participants meet inclusion criteria. Beck Depression Inventory II (BDI-II). The BDI-II is the third-generation BDI, revised in 1996, and based on the original. The instrument retains its original 21-item questionnaire format that requires approximately 10 min to complete. This indicator is used in the trials to monitor participants' mood during the study, making it also a measure for participants' safety. Participants will complete this measure during screening and daily during inpatient episodes. Visual Analogue Scales (VAS). Subjective effects produced by cocaine or placebo will be measured using a VAS consisting of a continuous 10-cm line marked from 0 to 100. Participants will be required to rate their drug craving, dysphoria, and euphoria on a scale from 0 to 100. Ratings include "High," "Good Effects," "Bad Effects," "Like Drug," "Dislike Drug," "Crave Cocaine," "Likely to Use Cocaine if Available", and "Desire Cocaine."

ELIGIBILITY:
Inclusion Criteria:

1. Be English-speaking volunteers who are not seeking treatment at the time of the study. We require proficiency in English to ensure good communication with staff
2. Be aged between 18 and 55 years
3. Meet DSM-IV TR criteria for cocaine dependence using the MINI
4. Have a self-reported history of using cocaine by the IV or smoked route
5. Have vital signs as follows: resting pulse between 50 and 95 bpm, BP between 90-150 mmHg systolic and 45-95 mmHg diastolic
6. Have hematology and chemistry laboratory tests that are within reference limits (±10%), with the following exceptions: (a) liver function tests (total bilirubin, ALT, AST, and alkaline phosphatase) <3× the upper limit of normal and (b) kidney function tests (creatinine and BUN) <2× the upper limit of normal
7. Have a baseline ECG that demonstrates clinically normal sinus rhythm, clinically normal conduction, and no clinically significant arrhythmias
8. Have a medical history and brief physical examination demonstrating no clinically significant contraindications for study participation, in the judgment of the admitting physician and the principal investigator

Exclusion Criteria:

1. Have any history or evidence suggestive of seizure disorder or brain injury
2. Have any previous medically adverse reaction to cocaine, including loss of consciousness, chest pain, or epileptic seizure
3. Meet criteria for current dependence on any drug other than cocaine or nicotine
4. Have neurological or psychiatric disorders, such as:

   * psychosis, bipolar illness or major depression as assessed by MINI;
   * organic brain disease or dementia assessed by clinical interview;
   * history of any psychiatric disorder that would require ongoing treatment or that would make study compliance difficult;
   * and history of suicide attempts within the past year and/or current suicidal ideation/plan
5. Have evidence of clinically significant heart disease or hypertension, as determined by the PI
6. Have a family history in first-degree relatives of early cardiovascular morbidity or mortality, as determined by the PI
7. Have evidence of untreated or unstable medical illness including neuroendocrine, autoimmune, renal, hepatic, or active infectious disease
8. Have HIV and are currently symptomatic or are taking antiretroviral medication
9. Be pregnant or nursing. Females must provide negative pregnancy urine tests upon hospital admission and at the end of study participation. Females must either be unable to conceive (i.e., surgically sterilized, sterile, or postmenopausal) or be using a reliable form of contraception (e.g., abstinence, birth control pills, intrauterine device, condoms, or spermicide)
10. Have asthma or currently use theophylline or other sympathomimetics
11. Be taking a medication that potently inhibits CYP 3A4, as this enzyme metabolizes the study medications. Potent inhibitors include clarithromycin, indinavir, itraconazole, ketoconazole, nefazodone, nelfinavir, ritonavir, saquinavir, telithromycin, or voriconazole
12. Have any other illness, condition, or use of psychotropic medications, which in the opinion of the PI and/or the admitting physician would preclude safe and/or successful completion of the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2018-08-21 (Actual); Study Completion 2018-08-21 (Actual)

PRIMARY OUTCOMES:
Subjective effects (VAS) - change from baseline over 60 minutes | baseline-post cocaine (5, 15, 30, 45, and 60 minutes following each infusion)
  difference between the peak "High" VAS rating observed post-cocaine infusion and that observed at baseline prior to the infusion

SECONDARY OUTCOMES:
heart rate change from baseline over 60 minutes | baseline-post cocaine (continuous first 30 minutes post cocaine session and 45 and 60 min post cocaine)
blood pressure change from baseline over 60 minutes | baseline-post cocaine (continuous first 30 minutes post cocaine session and 45 and 60 min post cocaine)

CONTACTS AND LOCATIONS:
Locations (1):
- Michael Debakey VA Medical Center, Houston, Texas, United States